CLINICAL TRIAL: NCT01770002
Title: Eversion in Dermatologic Surgery: Is Cosmetic Appearance Improved?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 265161
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma; Melanoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Melanoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everted suture technique (Active Comparator): Technique that everts the skin; the edges will sit up against each other in a little peak, raised above the surrounding skin.
  Interventions: Procedure: Everted suture technique
- Non-everted suture technique (Active Comparator): Surgical wound will be approximated such that the suture line is flat relative to the surrounding skin.
  Interventions: Procedure: Non-everted suture technique

INTERVENTIONS:
Procedure: Everted suture technique
  Arms: Everted suture technique
Procedure: Non-everted suture technique
  Arms: Non-everted suture technique

SUMMARY:
The investigators hypothesize that everting wound edges while suturing surgical sites will result in more aesthetic scars. Additionally, we also hypothesize that small to moderate wound irregularities present at 3 months will resolve by 6 months after surgery with no intervention

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to give informed consent themselves
* Willing to return for follow up visits

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Unwilling to return for follow up
* Pregnant Women
* Wounds less than 3 cm in length

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Everted versus non-everted suturing techniques | 3 and 6 months
  Primary outcome measures for this study are the post operative scar width measured at 1 cm from the midline on both sides of the scar.
Mean score of sum of 2 blinded observers POSAS scores | 3 and 6 months
  The mean summed total of two blinded reviewers Physician Observer Scar Assessment Scale (POSAS) scores for each side of the wound.
Scar measurements (height, width, length) | 3 and 6 months
  Scar volume will be measured in centimeters on both sides of the wound
Scar induration | 3 and 6 months
  Scar induration area will be measured in centimeters for both sides of the wound
Scar erythema | 3 and 6 months
  Scar erythema area will be measured in centimeters for both sides of the wound
Wound contour irregularities | 3 and 6 months
  Wound contour irregularities will be measured in terms of volume in cubic centimeters via a length, width and height measurement
Stand cone volume | 3 and 6 months
  The volume of standing cones will be measured via length, width and height measurements in centimeters
Uneven edge measurement | 3 and 6 months
  The area of uneven edges will be measured via a length x height measurement in centimeters
Hyperpigmentation area | 3 and 6 months
  areas of hyperpigmentation will be measured via a length x width measurement in centimeters

SECONDARY OUTCOMES:
Infection | up to 6 months
  Infections occurring anytime during the study period will be recorded
wound dehiscence | up to 6 months
  incidence of wound infection will be recorded anytime during the study period
spitting sutures | 3 and 6 months
  spitting sutures will be counted for each side of the wound at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical